CLINICAL TRIAL: NCT01210092
Title: Comparison of Different Video Laryngoscopes in a Manikin With Immobilized Cervical Spine
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, J. Hinkelbein, PD Dr. med., University of Cologne
Other Study IDs: 10-182-2
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Tracheal Intubation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Macintosh #3 Laryngoscope
- Glidescope
- Ambu Pentax AWS
- McGrath
- Airtraq
- Storz C-MAC

SUMMARY:
To determine whether different video laryngoscopes facilitate intubation in an manikin with immobilized cervical spine compared with standard laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* anaesthesiologist
* experienced in tracheal intubation

Exclusion Criteria:

* missing experience in tracheal intubation
* missing informed consent

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: anaesthesiologists
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
successful tracheal intubation | max 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang A Wetsch, MD, Principal Investigator — Department of Anaesthesiology, University of Cologne
Locations (1):
- Department of Anaesthesiology and Postoperative Critical Care, Cologne, Germany